CLINICAL TRIAL: NCT03846180
Title: Terlipressin Versus Somatostatin/Octreotide on Effect of Renal Function in Cirrhotic Patients With Acute Gastrointestinal Hemorrhage (TORCH): A Retrospective Multicenter Observational Study
Brief Title: Terlipressin on Effect of Renal Function in Cirrhotic Patients With Acute Gastrointestinal Hemorrhage
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Principal Investigator, General Hospital of Shenyang Military Region
Other Study IDs: XHNKKY-VASO 2.0
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Variceal Hemorrhage; Cirrhosis, Liver; Kidney Injury
MeSH Terms: conditions — Liver Cirrhosis | interventions — Terlipressin; Somatostatin; Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Terlipressin group: Cirrhotic patients with acute gastrointestinal bleeding received terlipressin with or without somatostatin/octreotide.
  Interventions: Drug: Terlipressin
- Somatostatin/Octreotide group: Cirrhotic patients with acute gastrointestinal bleeding received somatostatin and/or octreotide without terlipressin.
  Interventions: Drug: Somatostatin; Drug: Octreotide

INTERVENTIONS:
Drug: Terlipressin — Continuous or intermittent intravenous infusion of terlipressin was given.
  Other Names: Glypressin
  Groups: Terlipressin group
Drug: Somatostatin — Continuous or intermittent intravenous infusion of somatostatin was given.
  Other Names: Stilamin
  Groups: Somatostatin/Octreotide group
Drug: Octreotide — Continuous or intermittent intravenous infusion of octreotide was given.
  Other Names: Sandostatin
  Groups: Somatostatin/Octreotide group

SUMMARY:
Terlipressin and somatostatin/octreotide are the first-line choices for the treatment of acute variceal bleeding in liver cirrhosis. Acute kidney injury can develop in patients presenting with acute variceal bleeding. On the other hand, evidence suggests that terlipressin can reverse hepatorenal syndrome. It has been hypothesized that terlipressin can protect the renal function in cirrhotic patients with acute variceal bleeding, except for control of bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhotic patients who were admitted between January 2010 and December 2018.
2. A diagnosis of acute gastrointestinal bleeding.
3. Patients who received terlipressin or somatostatin/octreotide.
4. Age or sex was not limited.
5. Use of endoscopy was not limited.
6. Comorbidity was not limited.
7. Malignancy was not limited.

Exclusion Criteria:

1. Renal parenchymal diseases.
2. Absence of baseline serum creatinine.
3. Absence of serum creatinine 3-5 days after terlipressin or somatostatin/octreotide.
4. Duration of terlipressin or somatostatin/octreotide was less 3 days.
5. Patients who underwent transjugular intrahepatic portosystemic shunt.
6. Patients who underwent surgical shunt, splenectomy with or without devascularization, or liver transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cirrhotic patients with acute gastrointestinal bleeding received terlipressin or somatostatin/octreotide.
Sampling Method: Non-Probability Sample
Enrollment: 1682 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ICA-AKI and kidney function damage in cirrhotic patients with acute gastrointestinal bleeding | Through study completion, an average of 1-2 weeks
  ICA-AKI and kidney function damage
Effect of ICA-AKI and kidney function damage on in-hospital mortality of cirrhotic patients with acute gastrointestinal bleeding | Through study completion, an average of 1-2 weeks
  In-hospital mortality
Effect of terlipressin on the in-hospital mortality of cirrhotic patients with acute gastrointestinal bleeding with ICA-AKI and kidney function damage | Through study completion, an average of 1-2 weeks
  In-hospital mortality associated with ICA-AKI and kidney function damage

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Center for Liver Cirrhosis, The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Difficult & Complicated Liver Diseases and Artificial Liver Center, Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Liver Research Center, The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Department of Hepatobiliary Disease, 900 Hospital of the Joint Logistics Team (formerly called Fuzhou General Hospital), Fuzhou, Fujian
  - Department of Gastroenterology, The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Department of Gastroenterology, The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Department of Critical Care Medicine, The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Department of Gastroenterology, Air Force Hospital of Northern Theater Command, Shenyang, Liaoning
  - Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning
  - Department of Gastroenterology, Xi'an Central Hospital, Xi'an, Shaanxi
  - Department of Gastroenterology, Shandong Provincial Hospital Affiliated to Shandong University, Jinan, Shandong
  - Eastern Hepatobiliary Hospital of the Second Military Medical University, Shanghai, Shanghai Municipality
  - Department of Gastroenterology, General Hospital of Western Theater Command, Chengdu, Sichuan
  - State Key Laboratory for Diagnosis and Treatment of Infectious Diseases, Collaborative Innovation Center for Diagnosis and Treatment of Infectious Diseases, The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
This plan to share the individual patient data has been not decided yet.

REFERENCES:
- [Background] Zhang J, Rossle M, Zhou X, Deng J, Liu L, Qi X. Terlipressin for the treatment of hepatorenal syndrome: an overview of current evidence. Curr Med Res Opin. 2019 May;35(5):859-868. doi: 10.1080/03007995.2018.1552575. Epub 2019 Jan 4. PMID 30474439
- [Background] Zhou X, Tripathi D, Song T, Shao L, Han B, Zhu J, Han D, Liu F, Qi X. Terlipressin for the treatment of acute variceal bleeding: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Nov;97(48):e13437. doi: 10.1097/MD.0000000000013437. PMID 30508958
- [Background] Zhou XM, Qi XS, Jia JD. [An evidence-based terlipressin therapy for gastroesophageal variceal hemorrhage]. Zhonghua Gan Zang Bing Za Zhi. 2018 Apr 20;26(4):245-248. doi: 10.3760/cma.j.issn.1007-3418.2018.04.002. Chinese. PMID 29996332
- [Derived] Xu X, Liu B, Lin S, Li B, Wu Y, Li Y, Zhu Q, Yang Y, Tang S, Meng F, Chen Y, Yuan S, Shao L, Bernardi M, Yoshida EM, Qi X. Terlipressin May Decrease In-Hospital Mortality of Cirrhotic Patients with Acute Gastrointestinal Bleeding and Renal Dysfunction: A Retrospective Multicenter Observational Study. Adv Ther. 2020 Oct;37(10):4396-4413. doi: 10.1007/s12325-020-01466-z. Epub 2020 Aug 28. PMID 32860184